CLINICAL TRIAL: NCT00693160
Title: Effect of Intrathecal Ketorolac on Mechanical Hypersensitivity Following Acute Opioid Exposure
Brief Title: Effect of Spinal Ketorolac After Acute Opioid Exposure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the manufacturing of preservative free ketorolac (Acular-PF) was discontinued
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00002457; GM48085
Record Dates: First submitted 2008-02-15; First posted 2008-06-06 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: healthy volunteers; analgesia; pain; Healthy subjects
MeSH Terms: conditions — Agnosia; Pain | interventions — Ketorolac; Ketorolac Tromethamine; Remifentanil; Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intrathecal Ketorolac (Experimental): In the presence of a remifentanil infusion subject will receive a single intrathecal injection of ketorolac 2 mg Each subject will receive the topical capsaicin model for hyperalgesia and allodynia assessment.
  Interventions: Drug: ketorolac; Drug: remifentanil; Drug: Capsaicin
- Placebo intrathecal injection (Placebo Comparator): In the presence of remifentanil the subject will receive a single intrathecal injection of placebo (preservative-free normal saline) Each subject will receive the topical capsaicin model for hyperalgesia and allodynia assessment.
  Interventions: Drug: placebo; Drug: remifentanil; Drug: Capsaicin

INTERVENTIONS:
Drug: ketorolac — single intrathecal injection of ketorolac 2 mg
  Other Names: toradol; acular pf
  Arms: Intrathecal Ketorolac
Drug: placebo — subject will receive a placebo (preservative free normal saline) spinal injection
  Arms: Placebo intrathecal injection
Drug: remifentanil — All subjects will receive a remifentanil infusion
  Other Names: ultiva
Drug: Capsaicin — Topical capsaicin pain model utilized for each subject

SUMMARY:
This research study is being done because pain is a significant problem for patients with a variety of medical problems and following surgery or traumatic injury. Currently available pain medications may not treat all types of pain or may treat pain only at doses that produce side effects and complications. The medication in this study may have a role in better treatment of pain. The goals of this study are to see if a dose of ketorolac (non-narcotic, pain reliever), given into the fluid in the back near the spine has any effect on pain or discomfort in the skin sensation that will take place after applying capsaicin (chili pepper) cream. The sunburn-like sensation that people experience after having capsaicin cream applied is similar to, but much milder than, the pain that some people have after surgery and after certain types of nerve injuries. This study will test the effects of combining two medications that are often given together to control postoperative pain or pain from a nerve injury. The investigators are especially interested in answering two questions about the effects of ketorolac (non-narcotic pain reliever) and remifentanil (intravenous [IV] narcotic painkiller):

1. How much does remifentanil (narcotic painkiller) affect the sunburn-like painful area on your skin, which develops after applying capsaicin cream?
2. What pain relieving effects does spinal ketorolac have when given with IV remifentanil?

DETAILED DESCRIPTION:
Intravenous (IV) remifentanil stimulates spinal COX activity, leading to increased Cerebrospinal fluid CSF) prostaglandin E2 (PGE2) concentrations and areas of capsaicin-induced mechanical hypersensitivity after remifentanil infusion, and these effects will be blocked by intrathecal ketorolac.

Areas of mechanical hyperalgesia and allodynia will be established by topical capsaicin + intermittent heat in healthy volunteers, who will be randomized to receive intrathecal saline or ketorolac during remifentanil infusion, with primary outcome measure area of hyperalgesia and secondary outcome measure Cerebrospinal fluid (CSF) prostaglandin E2 (PGE2) concentration after stopping remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* American Society of Anesthesiologist (ASA) I or II classification
* between the ages of 18-55
* weigh less than 250 pounds
* without chronic pain

Exclusion Criteria:

* taking analgesics in the last 2 weeks
* positive urine drug screen
* pregnancy
* currently taking any prescription antidepressants or other medications that are mood altering
* liver or kidney disease
* stomach ulcers
* allergies to ketorolac, lidocaine, or capsaicin cream
* lung disease (COPD)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 healthy subjects between the ages of 19-51 were recruited and 30 were randomized between the dates for 11/20/2007 and 8/17/2010. Subjects were seen for all study related visits in the General Clinical Research Center at Wake Forest Baptist Medical Center in Winston-Salem, North Carolina.
Groups:
- Intrathecal Ketorolac: In the presence of a remifentanil infusion subjects received a single intrathecal injection of ketorolac 2 mg.
  The remifentanil infusion was initiated in each subject to a target concentration of 1.0 ng/ml using a computer controlled pump and the STANPUMP algorithm. The STANPUMP program, written by Dr. S.L. Shafer of Stanford University permits the administration of a pharmacokinetically tailored infusion to rapidly achieve and maintain a targeted plasma drug concentration.
  The remifentanil infusion was titrated based on the subjects' pain report to a 49 degree Celsius stimulus with the goal of producing approximately 50% decrease in verbal pain report of the 49 degree Celsius stimulus. Upon reaching the target concentration, a steady state infusion was then completed over 80-to 100 minutes.
- Placebo Intrathecal Injection: In the presence of remifentanil subjects received a single intrathecal injection of placebo (preservative-free normal saline).
  The remifentanil infusion was initiated in each subject to a target concentration of 1.0 ng/ml using a computer controlled pump and the STANPUMP algorithm. The STANPUMP program, written by Dr. S.L. Shafer of Stanford University permits the administration of a pharmacokinetically tailored infusion to rapidly achieve and maintain a targeted plasma drug concentration.
  The remifentanil infusion was titrated based on the subjects' pain report to a 49 degree Celsius stimulus with the goal of producing approximately 50% decrease in verbal pain report of the 49 degree Celsius stimulus. Upon reaching the target concentration, a steady state infusion was then completed over 80-to 100 minutes.
Period: Overall Study
Arm/Group | Intrathecal Ketorolac | Placebo Intrathecal Injection
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intrathecal Ketorolac: In the presence of a remifentanil infusion subject will receive a single intrathecal injection of ketorolac 2 mg
- Placebo Intrathecal Injection: In the presence of remifentanil the subject will receive a single intrathecal injection of placebo (preservative-free normal saline)
- Total: Total of all reporting groups
Arm/Group | Intrathecal Ketorolac | Placebo Intrathecal Injection | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.78 (11.52) | 32.06 (8.52) | 31.93 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hyperalgesia
Description: Total Area of hypersensitivity (measured in centimeters) were assessed approximately 24 hours post intrathecal ketorolac injection by the method of using a von Frey filament
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: centimeters^2
Arm/Group | Intrathecal Ketorolac | Placebo Intrathecal Injection
Number analyzed (Participants) | 14 | 16
centimeters^2 | 70.1 (40.5) | 48.4 (33.5)

2. Secondary Outcome: Cerebrospinal Fluid (CSF) Prostaglandin E2 (PGE2) Concentration
Description: Concentration of prostaglandin E2 (PGE2) in Cerebrospinal fluid (CSF) 2.5 hours post injection of intrathecal ketorolac
Time Frame: 2.5 hours
Population: 11 Subjects in the Intrathecal Ketorolac group received post study treatment analysis of CSF for PGE2. We were not able to obtain CSF samples in 3 of the subjects post study drug injection.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Intrathecal Ketorolac | Placebo Intrathecal Injection
Number analyzed (Participants) | 11 | 16
picograms per milliliter | 87 (95) | 75 (41)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Subjects were followed up for 2 weeks and questioned for any adverse events
Arm/Group | Intrathecal Ketorolac | Placebo Intrathecal Injection
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes